CLINICAL TRIAL: NCT06465368
Title: AN INTERVENTIONAL, OPEN-LABEL, RANDOMIZED, MULTICENTER, PHASE 2 STUDY OF PF-07220060 PLUS LETROZOLE COMPARED TO LETROZOLE ALONE IN POSTMENOPAUSAL WOMEN 18 YEARS OR OLDER WITH HORMONE RECEPTOR-POSITIVE, HER2-NEGATIVE BREAST CANCER IN THE NEOADJUVANT SETTING
Brief Title: A Study to Learn About the Study Medicine PF-07220060 Together With Letrozole Compared to Letrozole Alone in Women Post Menopause
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4391025; 2024-512848-30-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: human epidermal growth factor receptor 2 (HER2); hormone receptor (HR); HER2-negative; HR-Positive; Breast Cancer (BC); Neoadjuvant; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A/Experimental/PF-07220060 plus letrozole (Experimental): PF-07220060 given as tablet by mouth twice a day for 14 days. Letrozole given as tablet by mouth once a day for 14 days.
  Interventions: Drug: PF-07220060; Drug: letrozole
- Arm B/Control/letrozole (Active Comparator): Letrozole given by mouth once a day for 14 days.
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: PF-07220060 — PF-07220060 given as tablet by mouth twice a day for 14 days.
  Arms: Arm A/Experimental/PF-07220060 plus letrozole
Drug: letrozole — Letrozole given as tablet by mouth once a day for 14 days
  Other Names: Femara

SUMMARY:
The purpose of this study is to learn about the effects of the study medicine PF-07220060 plus letrozole, compared with the effects of taking letrozole alone without PF-07220060 for treatment of breast cancer.

This study is seeking for participants who are:

* women of age 18 years and older post menopause (either naturally or surgically).
* confirmed to have Hormone receptor (HR) positive, Human epidermal growth factor receptor 2 (HER2) negative breast cancer. HER2 negative describes cells that have a small amount or none of a protein called HER2 on their surface. In normal cells, HER2 helps control cell growth. Cancer cells that are HER2 negative may grow more slowly and are less likely to recur (come back) or spread to other parts of the body than cancer cells that have a large amount of HER2 on their surface.
* not been treated for their cancer before this study.

Participants will be randomly assigned (like flipping a coin) to receive the treatment (PF-07220060 plus letrozole) or letrozole alone. Both PF-07220060 and letrozole are taken by mouth. PF-07220060 will be taken twice a day for 14 days. Letrozole will be taken once a day for 14 days.

Participants will have a screening period for up to 28 days. If deemed fit, they will receive study treatment for 14 days, and then will have a follow-up visit about 28 days after their last dose.

All participants will have at least one biopsy during the study. Biopsy is the removal of cells or tissues for examining. All participants will have a biopsy on Day 14.

Additional assessments for safety including blood draws and interviews done by the site staff will be completed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with histologically confirmed HR-positive and HER2-negative BC (per local assessment)
* Documented by estrogen receptor (ER) and/or progesterone receptor (PR)-positive disease by IHC or ISH
* Participants must have Ki-67 score >/=10% with unilateral, invasive T1c-T4c, N0-N2, M0 BC
* Participants must be willing and able to undergo a baseline and Day 14 biopsy and must have an ECOG PS or 0 or 1.
* Participants must be treatment naive for the treatment of BC and cannot have had prior treatment with any systemic therapy (e.g., chemotherapy, hormonal therapy), radiation, surgery, or any investigational agents or use of hormone replacement therapy (HRT) or any other estrogen-containing medication (including vaginal estrogen) within 2 weeks prior to diagnostic tissue sample taken.

Exclusion Criteria:

* No prior systemic therapy, radiation, surgery, investigational therapy for treatment of breast cancer
* Certain medical conditions in the previous 6 months, for example: myocardial infarction, severe unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association class III or IV), cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism or other clinically significant episode of thromboembolism
* Lab abnormalities outside protocol specified parameters

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 121 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Rate of Ki-67 | Day 14
  Centrally assessed biopsy

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Baseline, Day 14, and Day 28 post last treatment follow-up visit
Incidence of Serious AEs | Baseline, Day 14, and Day 28 post last treatment follow-up visit
Incidence of AEs leading to Discontinuation | Baseline, Day 14, and Day 28 post last treatment follow-up visit
Ctrough and peri-biopsy plasma concentrations of PF-07220060 | Pre-dose within 30 minutes and post-dose within 1 hour before or after biopsy
  Ctrough was defined as pre-dose serum concentration during multiple dosing and observed directly from data.
Circulating tumor DNA (ctDNA) measurements | Baseline and Day 14
  Evaluate response on treatment
Percentage of Ki-67 | Screening and Day 14
  All participants will have Ki-67 staining from the biopsy sample on Day 14 and Screening if not previously available

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (10):
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - AMG -Crystal Lake, Crystal Lake, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Advocate Medical Group, Park Ridge, Illinois
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas
  - O'Quinn Medical Tower - McNair Campus, Houston, Texas
  - START San Antonio, San Antonio, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (2):
  - Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de
  - UZ Leuven, Leuven, Vlaams-brabant
- France (7):
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer, Rennes, Ille-et-vilaine
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-roussillon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-atlantique
  - CHU de Saint-Etienne, Saint Priest En Jarez, Pays de la Loire Region
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - HCL, Centre Hospitalier Lyon Sud, Saint-Genis-Laval, Rhône
  - Gustave Roussy, Villejuif, Val-de-marne
- CaritasKlinikum Saarbrücken St. Theresia, Saarbrücken, Saarland, Germany
- Italy (5):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Azienda USL Toscana Nord Ovest_Ospedale Civile di Livorno, Livorno, Tuscany
  - Ospedale Antonio Perrino, Brindisi
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
- Poland (4):
  - AIDPORT Sp. z o.o., Skórzewo, Greater Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl, Podkarpackie Voivodeship
- Slovakia (2):
  - Nemocnica AGEL Komarno, Komárno, Nitra Region
  - Narodny onkologicky ustav, Bratislava
- Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul], South Korea
- Spain (10):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Región de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario HM Sanchinarro, Madrid
- Sweden (2):
  - Sjukhuset I Gävle, Gävle, Gävleborgs LÄN [se-21]
  - Akademiska sjukhuset, Uppsala, Uppsala LÄN [se-03]
- Switzerland (3):
  - Tumor Zentrum Aarau, Aarau, Canton of Aargau
  - University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Baden, Baden
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391025